CLINICAL TRIAL: NCT04349163
Title: Resilience Evaluation of Caregivers During the SARS-CoV2 Epidemic Period
Brief Title: Resilience Evaluation of Caregivers During the SARS-CoV2 Epidemic Period : Prospective Cohort.
Acronym: Resi-CoV
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-A00831-39
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-05

CONDITIONS: Psychological
Keywords: caregivers; covid-19; resilience; questionnaire; CD-RISC 25
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers: Physicians and nurses working at the Emergency Department, Intensive care Unit, infectious disease Department, Anaesthesiology.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — CD-RISC 25 questionnaire

SUMMARY:
The outbreak linked to SARS-CoV-2 infection was declared a Public Health Emergency of International Concern on 30 January 2020. In all of the emergency Departments, a major reorganization was necessary, notably with the creation of a specific channel for COVID-19 suspect patients. Thus, all caregivers involved must adapt day by day to new places of exercise, new protocols,...The major influx of patients, the precautions to be taken, the specifics of the pathology and its management have profoundly changed daily practice. This exogenous hospital tension impacts all caregivers and more particularly their resilience capacities. Resilience is defined as an ability to recover from or adjust easily to misfortune or change. The Resi-CoV study aims to assess the level of resilience of caregivers of different specialties and trades in the context of covid-19.

DETAILED DESCRIPTION:
Caregivers will be invited to complete a self-administered questionnaire online via a personalized electronic message. Caregivers will be free to participate. Signed consent will not be requested, but the return of the questionnaire will be considered consent. The questionnaire will be administered using Google form® software. Caregivers will have 2 weeks to respond. A reminder will be made at 7 days. The questionnaire will be anonymized upon receipt by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers (physicians, nurses)
* working in the Emergency Department, Anaesthesiology, Infectious Department, Intensive care Unit.
* Voluntary to answer the questionnaire

Exclusion Criteria:

- Working in another Department

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All caregivers willing to answer.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
compare the level of resilience between physicians and caregivers of different specialties and in different workplaces according to the covid-19 epidemic. | 14 days
  CD-RISC-25 : Connor-Davidson Resilience Scale - 25. This scale contain 25 questions each range from 1 to 5. The total is 100 points which means a very high level of resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Douillet, Principal Investigator — UH Angers
Locations (1):
- CHU, Angers, France